CLINICAL TRIAL: NCT06104553
Title: A Phase Ib/II Study of SHR-A1912 Combined With Other Therapies in Patients With B-cell Non-Hodgkin 's Lymphoma
Brief Title: A Trial of SHR-A1912 Combined With Other Therapies in B-cell Non-Hodgkin 's Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1912-II-201
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: An open, multicenter, dose-finding and dose expansion investigational Phase Ib/II clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1912 combined with R-Chemo (Phase 1b) (Experimental)
  Interventions: Drug: SHR-A1912; R-Chemo
- SHR-A1912 combined with R-Chemo (Phase 2) (Experimental)
  Interventions: Drug: SHR-A1912; R-Chemo

INTERVENTIONS:
Drug: SHR-A1912; R-Chemo — SHR-A1912 combined with R-Chemo: SHR-A1912 + R-Chemo (Rituximab + Chemotherapy) (Phase 1b)
  Arms: SHR-A1912 combined with R-Chemo (Phase 1b)
Drug: SHR-A1912; R-Chemo — SHR-A1912 combined with R-Chemo: SHR-A1912 (RP2D) + R-Chemo (Rituximab + Chemotherapy) (Phase 2)
  Arms: SHR-A1912 combined with R-Chemo (Phase 2)

SUMMARY:
This study aims to evaluate the safety, PK and preliminary anti-tumour activity of SHR-A1912 combined with other therapies in patients with B-cell non-Hodgkin 's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to18 years old;
2. Eastern Cooperative Oncology Group (ECOG) performance status is 0 to 1;
3. Life expectancy >3 months;
4. Histologically confirmed B-cell B-cell non-Hodgkin's lymphoma;
5. Previous systematic anti-tumor therapy should meet the following requirements: 1) Relapsed and/or refractory disease after at least one (≥ 1) line of prior systemic therapy (relapsed/refractory cohort); 2) Previously untreated (naïve cohort).
6. At least one measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or one measurable extra nodal lesion, defined as > 1.0 cm in its longest diameter.

Exclusion Criteria:

1. Received autologous stem cell transplantation within 12 weeks before the first study treatment; previously received allogeneic stem cell transplantation; received Car-T cell therapy within 12 weeks before the first study treatment;
2. History of recent major surgery or severe trauma within 4 weeks before the first study treatment;
3. Received anti-tumour treatment within 2 weeks before the first study treatment;
4. Central nervous system (CNS) infiltration;
5. Active infection with HBV or HCV;
6. History of immunodeficiency, including HIV serotest positive, or other acquired or congenital immunodeficiency diseases, and active tuberculosis;
7. Active infection or unexplained fever>38.5℃;
8. History of severe cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: RP2D (Recommended Phase II Dose) of SHR-A1912 combined with immunochemotherapy | The RP2D for Phase 2 will be selected at the end of Phase 1b, approximately 12 months
Phase 1b: Incidence and severity of AE | Up to follow-up period, approximately 24 months]
Phase 2: Objective response rate | assessed up to approximately 24 months

SECONDARY OUTCOMES:
Phase 1b: Objective response rate | assessed up to approximately 24 months
Phase 1b: Complete response rate (CRR) | assessed up to approximately 24 months
Phase 1b: Duration of remission (DoR) | assessed up to approximately 24 months
Phase 1b: Progression-free survival (PFS) | assessed up to approximately 24 months
Phase 1b: Toxin binding antibody to SHR-A1912 | Up to follow-up period, approximately 24 months
Phase 1b: Total antibody to SHR-A1912 | Up to follow-up period, approximately 24 months
Phase 1b: Concentration of free toxin | Up to follow-up period, approximately 24 months
Phase 1b: Anti-drug antibodies (ADA) to SHR-A1912 | Up to follow-up period, approximately 24 months
Phase 2: Complete response rate (CRR) | assessed up to approximately 24 months
Phase 2: Duration of remission (DoR) | assessed up to approximately 24 months
Phase 2: Progression-free survival (PFS) | assessed up to approximately 24 months
Phase 2: Incidence and severity of AE | Up to follow-up period, approximately 24 months
Phase 2: Toxin binding antibody to SHR-A1912 | Up to follow-up period, approximately 24 months
Phase 2: Total antibody to SHR-A1912 | Up to follow-up period, approximately 24 months
Phase 2: Concentration of free toxin | Up to follow-up period, approximately 24 months
Phase 2: Anti-drug antibodies (ADA) to SHR-A1912 | Up to follow-up period, approximately 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided